CLINICAL TRIAL: NCT06837818
Title: To Explore the Optimal Dose of Dexmedetomidine for Skull Pin Fixation in Intracranial Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20250016
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Procedural Pain
Keywords: Skull pin fixation; dexmedetomidine; Target-controlled infusion
MeSH Terms: conditions — Pain, Procedural | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): skull pin fixation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The first patient was started on dexmedetomidine Cp 0.4 ng/ml, 2 minutes before the procedure, and the up and down method was used, with the Cp of dexmedetomidine adjusted to 0.05 ng/ml each time. The analgesia nociception index (ANI) during skull pin fixation is lower than (<) 30 and the heart rate (HR) and arterial blood pressure (ABP) exceed (>) 20% of the baseline (or the HR is >100 bpm and the ABP is >180/100 mmHg), indicating insufficient analgesia or hemodynamics (failure). If the patient is failure for the procedure, increase the Cp by 0.05 ng/ml for the next patient; the ANI is higher than or equal to (≥30) and the HR and ABP do not exceed 20% of the baseline or the HR is ≤100 bpm and the ABP is ≤180 /100 mmHg) indicates that the analgesia and hemodynamic stability are acceptable (success), and the next patient will be adjusted downward by 0.05 ng/ml.

SUMMARY:
Skull pin fixation is commonly used in intracranial surgery, which can increase the surgical field of view. Because skull pin fixation is a very irritating and painful medical treatment, it often results in tachycardia (>150-160 beats per min, bpm) and high blood pressure (BP) (>200/120 mmHg). Many strategies to reduce this painful stimulation include oral gabapentin, local injection of local anesthetics, scalp nerve blockade, and deepening the depth of anesthesia. Oral gabapentin must take 2 hr before surgery with many adverse effects such as nausea and vomiting. Local injection of local anesthetics and scalp nerve blockade require injections by neurosurgeons. Due to the manpower and time constraints, neurosurgeons cannot perform the two techniques. Therefore, it depends on anesthesiologists to prescribe more anesthetics to attenuate this intensity painful stimulation. Usually anesthesiologists will give propofol, opioids (fentanyl, alfentanil or remifentanil), α2 agonist (dexmedetomidine or clonidine), add inhalation anesthetics (sevoflurane or desflurane), and finally even use b-blocker to reduce hemodynamic instability (hyperdynamics).

Dexmedetomidine mainly produces a sedative effect by activating α2 adrenergic receptors in the central nervous system. Its α2:α1 ratio is 1620:1, showing high affinity for α2 receptors. Unlike other hypnotic drugs during death, dexmedetomidine keeps the patient in an awakenable state and does not affect respiratory function during sedation. Therefore, general anesthesia can be enhanced, providing sedation and analgesia and improving sleep quality.

Target-controlled infusion (TCI) pump systems can automatically adjust drug infusion rates based on the patient's weight, age, and other physiological parameters to achieve more precise drug concentrations. It can maintain a stable drug concentration and reduce the impact of drug fluctuations on patients, especially when long-term anesthesia or sedation is required. Therefore, using a TCI pump system to administer dexmedetomidine can ensure that the concentration we want can be accurately achieved when performing skull pin fixation. Our hospital has routinely used the Dyck mode of the TCI pump system to infuse dexmedetomidine 0.2-0.4 ng/ml during intracranial surgery.

In view of this, we wanted to observe patients undergoing intracranial surgery with skull pin fixation using the Dyck mode by the TCI pump system under the monitoring of analgesic nociceptive index and hemodynamics. In order to find out the most appropriate dexmedetomidine concentration during skull pin fixation to reduce hemodynamic fluctuations and insufficient pain management as a basis for future anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old and less than 80 years old, with ASA I~III. Patients who are expected to undergo intracranial surgery for skull pin fixation.

Exclusion Criteria:

* Patients under the age of 18, patients over 80, those who have not signed a consent form, those with ASA class IV or higher, those who are allergic to dexmedetomidine or propofol or remifentanil, sever bradycardia (HR<40 bpm), hypotension (<90/60 mmHg) and hypertension crisis (180/110 mmHg), and emergency patients, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
50% effect concentration of dexmedetomidine | up to 15 minutes (peri-fixation period)
  50% effect concentration of dexmedetomidine will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.
95% effect concentration of dexmedetomidine | up to 15 minutes (peri-fixation period)
  95% effect concentration of dexmedetomidine will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.